CLINICAL TRIAL: NCT01077570
Title: The Clinical Safety and Effectiveness of Repaglinide in Treatment-naive Type 2 Diabetes Subjects in China. A 16-week Multicentre, Prospective, Open Label, Non-interventional Study.
Brief Title: An Observational Study Investigating the Safety and Effectiveness of Repaglinide in Chinese Patients
Acronym: SAFE
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: AGEE-3822; U1111-1112-6394 (Other: WHO)
Record Dates: First submitted 2010-02-26; First posted 2010-03-01 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — repaglinide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Repaglinide
  Interventions: Drug: repaglinide

INTERVENTIONS:
Drug: repaglinide — Repaglinide prescribed at the discretion of the investigator, according to local labelling, and evaluated at week 0, 8 and 16 of the study

SUMMARY:
This study is conducted in Asia. The aim of this observational study is, under normal clinical practice conditions, to investigate the clinical safety and effectiveness in Chinese patients with type 2 diabetes who have never received anti-diabetic treatment before.

ELIGIBILITY:
Inclusion Criteria:

* HbA1c more than 6.5%, no anti-diabetes treatment accepted before entering the study

Exclusion Criteria:

* Subjects who received any anti-diabetic treatment previously
* Known or suspected allergy to trial product(s) or related products.
* Subjects who previously enrolled in this study.
* Females of childbearing potential who are pregnant, breast-feeding or intend to become pregnant or are not using adequate contraceptive methods.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from both general and speciality practice settings who have been deemed appropriate to receive Repaglinide as initial treatment and as part of routine out-patient care by the prescribing physician.
Sampling Method: Non-Probability Sample
Enrollment: 2033 (Actual)
Dates: Start 2010-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Number of serious adverse drug reactions (SADRs) including major hypoglycaemic (low blood sugar) events | at Visit 2(8 weeks) and visit 3(16 weeks)

SECONDARY OUTCOMES:
Number of minor hypoglycaemic (low blood sugar) episodes | at Visit 2(8 weeks) and visit 3(16 weeks)
Number of adverse drug reactions (ADRs) | at Visit 2(8 weeks) and visit 3(16 weeks)
Change in HbA1c | after 16 weeks of treatment
Change in fasting blood glucose (FBG) | after 8 and 16 weeks of treatment
Change in postprandial blood glucose (PBG) | after 8 and 16 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Beijing, Beijing Municipality, China

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com